CLINICAL TRIAL: NCT04225897
Title: A Phase 2 Open-Label Study in Infants With REspiratory Syncytial VIRus Lower RespirAtory Tract Infection, Followed by a DoubLe-blind, Placebocontrolled Part, to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Effect of RV521 (REVIRAL 1)
Brief Title: A Study to Learn About the Effects of Sisunatovir in Infants With Respiratory Syncytial Virus Lower Respiratory Tract Infection.
Acronym: REVIRAL 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Part A and Part B were completed but Pfizer terminated Part C due to strategic consideration. There were no safety concerns in the decision to stop Part C and no changes to the risk-benefit for participants who received RV521 in the study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: REVC003; C5241003 (Other: Alias Study Number)
Record Dates: First submitted 2019-12-11; First posted 2020-01-13 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Syncytial Virus (RSV); Lower Resp Tract Infection
Keywords: RV521; Pediatrics; Children; LRTI; Wheezing; Rhinitis; Cough; sisunatovir
MeSH Terms: conditions — Respiratory Sounds; Rhinitis; Cough | interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: This is a multicentre, 3-part study to evaluate safety, tolerability, PK, PD, and antiviral effect of single and multiple dosing of RV521 in infants hospitalised due to RSV LRTI. Due to the adaptive study design, the number of enrolled subjects may vary depending on the obtained PK and safety profiles.
  The clinical study consists of 3 parts:
  * Part A is an open-label, multicentre, single dose study in infants hospitalised with RSV LRTI (Cohorts 1 & 2)
  * Part B is a randomised, double-blind, placebo-controlled, multicentre multiple dose study in infants hospitalised with RSV LRTI (Cohorts 3, 4 & 5)
  * Part C is a randomised 1:1, double-blind, placebo-controlled, multicentre, multiple-dose study in infants hospitalised with RSV LRTI
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RV521 (Experimental): sisunatovir is formulated as a dry powder blend of RV521 drug substance with mannitol as excipient. The RV521 dry powder blend will be supplied in capsules containing 10, 20, or 50 mg RV521. The Investigational Medicinal Product (IMP) will be dispersed in a defined volume of suspending diluent prior to oral administration on a mg/kg basis. Instructions for opening the capsule(s) and dispersing the contents in a fixed volume of suspending diluent prior to administration will be provided in the Pharmacy Manual.
  The proposed dosing regimen for Part A is a single open label dose of RV521. Part B and C is RV521 or placebo administered BID, 12 hours apart, for a period of 5 consecutive days with a total of 10 doses. However, this is subject to the recommendation of the DSMC.
  Interventions: Drug: RV521
- Placebo (Placebo Comparator): The placebo capsules administered in Part B and C will contain mannitol and microcrystalline cellulose (vehicle). The placebo dry powder will be dispersed in suspending diluent and given orally BID. Instructions for opening the capsule(s) and dispersing the contents in a fixed volume of suspending diluent prior to administration will be provided in the Pharmacy Manual.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV521 — RV521 is an RSV F protein inhibitor administered orally
  Other Names: sisunatovir
  Arms: RV521
Drug: Placebo — vehicle administered orally
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (sisunatovir). Sisunatovir is developed as potential treatment of Respiratory Syncytial Virus (RSV) infections. This study will assess sisunatovir as compared to placebo in infants aged 1 month to 36 months who are hospitalized with RSV lower respiratory tract infection (LRTI). A placebo looks like the study medicine but does not contain any active medicine in it.

This study will be conducted in 3 parts:

In Part A participants aged 6 months to 3 years will be given a single dose of 2.5 mg/kg of sisunatovir in Cohort 1. In Cohort 2, participants age 1 month to 6 months will receive a single dose of 2 mg/kg of sisunatovir only after the completion of Cohort 1. 12-24 participants will be enrolled in Part A In Part B participants age 1 month to 36 months will receive sisunatovir or placebo dosed every 12 hours for 5 days. Doses for part B will be determined after the completion of Part A. 24-40 participants will be enrolled in Part B.

The dose regimen for Part C will be determined after the completion of Part B. Approximately 120 participants age 1 month to 36 months will receive either sisunatovir or placebo.

To participate in this study participants must meet the following criteria:

1. Age 1 month to 36 months
2. Weight ≥ 3.5 kg
3. Diagnosis of LRTI
4. Diagnosis of RSV
5. Hospitalization due to RSV LRTI

DETAILED DESCRIPTION:
This is a multicentre, 3-part study to evaluate safety, tolerability, PK, PD, and antiviral effect of single and multiple dosing of RV521 in infants hospitalised due to RSV LRTI.

The clinical study consists of 3 parts, the third part (Part C) is optional:

* Part A is an open-label, multicentre, single dose study in infants hospitalised with RSV LRTI (Cohorts 1 & 2)
* Part B is a randomised, double-blind, placebo-controlled, multicentre multiple dose study in infants hospitalised with RSV LRTI (Cohorts 3, 4 & 5)
* Part C is a randomised 1:1, double-blind, placebo-controlled, multicentre, multiple-dose study in infants hospitalised with RSV LRTI I The number of subjects enrolled in Parts A and B of the study will depend on the safety and PK data from the group of subjects enrolled in specified age cohorts and the subsequent recommendation of the Data Safety Monitoring Committee (DSMC).

The DSMC may recommend a dose adjustment (either a reduction or an escalation) and/or regimen adjustment (Part B only) for subsequent subjects because of the observation of an unexpected safety/tolerability profile and/or differences between the observed and predicted exposure resulting from a specified dose of RV521.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 1 month and ≤ 36 months of age
2. Weight ≥ 3.5 kg
3. Clinical diagnosis of LRTI
4. A positive RSV diagnostic test
5. Hospitalised because of RSV LRTI
6. Symptoms of LRTI must be present for no more than 1 week (Part B) and no more than 5 days (Part C) before the Screening Visit
7. Expected to remain in hospital for a minimum of 3 days
8. The parent(s)/legal guardian(s) of the subject have provided written informed consent for the subject to participate and are able and willing to comply with the study protocol

Exclusion Criteria:

1. Premature (gestational age less than 37 weeks) AND <1 year of post-natal age
2. Known to have significant comorbidities that would limit the ability to administer study drug or evaluate the safety or clinical response to study drug.
3. Any clinically significant ECG abnormalities.
4. Known to be immunocompromised.
5. High risk of having developing asthma.
6. Suspected of having a clinically significant bacterial infection.
7. History of renal failure.
8. Clinical evidence of hepatic decompensation
9. History of epilepsy or seizures, including febrile seizures
10. Allergy to test medication or constituents
11. Has received 1 or more doses of palivizumab at any time before Screening or received treatment with antiviral therapy for RSV (eg, ribavirin or intravenous [IV] immunoglobulin) within 3 months before the Screening Visit.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Argentina (3):
  - Hospital Interzonal General de Agudos "Dr. José Penna", Bahía Blanca, Buenos Aires
  - Hospital Italiano Regional Del Sur, Bahía Blanca, Buenos Aires
  - Hospital General de Ninos Pedro de Elizalde, Buenos Aires, Buenos Aires F.D.
- Hospital de ninos "Ricardo Gutierrez", Calgary, Alberta, Canada
- Chile (2):
  - Hospital Base San Jose Osorno, Osorno, Los Lagos Region
  - Hospital de Ninos Dr. Roberto del Rio, Santiago, Santiago Metropolitan
- Costa Rica (5):
  - Corporacion Gihema, San José
  - Hospital Clinica Biblica, San José
  - Hospital Metropolitano, Sede San Jose, San José
  - lnstituto de lnvestigacion en Ciencias Medicas(IICIMED), San José
  - Policlinico San Bosco, Consultorio de Pediatria, Dr. Arturo Solis Moya, San José
- Hungary (3):
  - Semmelweis Egyetem 11.sz. Gyermeklinika, Budapest
  - Eszak-Kozep-budai Centrum,Uj Szent Janos Korhaz es Szakrendelo,Gyermekosztaly, Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Schneider Children's Medical Center of Israel, Petach Tikava
- Malaysia (7):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Taiping, Taiping, Perak
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - Hospital Seri Manjung, Parek
- Capital and Coast DHB, Wellington Hospital, Riddiford Street, Wellington Region, New Zealand
- Panama (3):
  - Hospital de Especialidades Pediatricas "Omar Torrijos Herrera", Panama City
  - Hospital del Nino Dr. Jose Renan Esquivel, Panama City
  - Hospital Materno Infantil Jose Domingo de Obaldia, Panama City
- Poland (3):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - lnstytut Centrum Zdrowia Matki Polki Klinika Pediatrii, Immunologii i Nefrologii, Lodz
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny w Warszawie Oddzial Kliniczny Pediatrii, Warsaw
- South Korea (2):
  - Seoul National University Children's Hospital, Seoul
  - Department of Pediatrics, SoonchunHyang University Seoul Hospital, Seoul
- Spain (9):
  - Hospital Universitario Sant Joan de Deu, Espluges de Llobregat, Barcelona
  - Fundacion Hospital de Nens, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Clinico de San carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Paz ,Pediatric Deparment, Madrid
  - Hospital Universitario La Paz Servicio de Farmacia. Planta baja Edificio Norte, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Santiago, Santiago de Compostela
- Taiwan (4):
  - Hsinchu Mackay Memorial Hospital, Hsinchu
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chi Mei Medical Center, Tainan
- Thailand (10):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - The Pharmacy Unit Ground Floor, OPD Building Faculty of Madicine,, Bangkoknoi, Bangkok
  - Chula Clinical Research Center, Faculty of Medicine, Patumwan, Bangkok
  - King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Bangkok
  - QueenSirikit National Institute of Child Health {QSNICH}, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital,Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiangrai
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Naresuan University Hospital ,Faculty of Medicine, Naresuan University, Phitsanulok
- United Kingdom (4):
  - Alder Hey Children's NHS Foundation Trust Institute in the Park, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust Evelina London Children's Hospital Westminster, London
  - Imperial College Healthcare NHS Trust St Mary's Hospital, London
  - University Hospital Southampton NHS Foundation Trust NIHR Clinical Research Facility ,Mailpoint 218,, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVC003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to be conducted in 3 parts: Part A, B and optional part C. Part C was not conducted as part of a reassessment of the clinical development plan for RV521 (sisunatovir); hence, data is not reported for Part C in any section of the results. A total of 51 participants were enrolled in the study (Part A=19 and Part B=32).
Groups:
- Cohort 1: RV521 1.0 mg/kg: Infants aged >=6 months to <=36 months hospitalized with respiratory syncytial virus lower respiratory tract infection (RSV LRTI) received a single dose of 1.0 milligram per kilogram (mg/kg) of RV521 orally on Day 1.
- Cohort 1: RV521 2.0 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 2.0 mg/kg of RV521 orally on Day 1.
- Cohort 1: RV521 2.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 2.5 mg/kg of RV521 orally on Day 1.
- Cohort 2: RV521 2.0 mg/kg: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received a single dose of 2 mg/kg of RV521 orally on Day 1.
- Cohort 3: Placebo: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received placebo every 12 hours twice daily (BID) orally for 5 days.
- Cohort 3: RSV1 2.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 2.5 mg/kg every 12 hours (BID) orally for 5 days.
- Cohort 3: RV521 3.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 3.5 mg/kg every 12 hours (BID) orally for 5 days.
- Cohort 3: RV521 5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 5 mg/kg every 12 hours (BID) orally for 5 days.
- Cohort 4: Placebo; Cohort 5: Placebo: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received placebo every 12 hours (BID) orally for 5 days.
- Cohort 4: RV521 2.5 mg/kg; Cohort 5: RV521 2.5 mg/kg: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received RV521 2.5 mg/kg every 12 hours (BID) orally for 5 days.
Period: Part A (Screening Visit to Day 7)
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Started | 3 | 7 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 3 | 7 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 6 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Parent/legal guardian request | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Screening Visit to Day 12)
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Started | 0 (No participants in Part B.) | 0 (No participants in Part B.) | 0 (No participants in Part B.) | 0 (No participants in Part B.) | 3 (Participants enrolled in Part B of the study.) | 3 (Participants enrolled in Part B of the study.) | 4 (Participants enrolled in Part B of the study.) | 3 (Participants enrolled in Part B of the study.) | 1 (Participants enrolled in Part B of the study.) | 4 (Participants enrolled in Part B of the study.) | 6 (Participants enrolled in Part B of the study.) | 8 (Participants enrolled in Part B of the study.)
Treated | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 3 | 1 | 4 | 6 | 8
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 2 | 1 | 4 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Parent/legal guardian request | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Cohort 1: RV521 1.0 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 1.0 milligram per kilogram (mg/kg) of RV521 orally on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg | Total
Number analyzed (Participants) | 3 | 7 | 3 | 6 | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8 | 50
Age, Customized [Count of Participants; unit: Participants]
  28 days to 23 months | 1 | 5 | 3 | 6 | 3 | 3 | 2 | 1 | 1 | 4 | 5 | 8 | 42
  2 to 11 years | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 2 | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 5 | 19
  Male | 3 | 3 | 1 | 5 | 2 | 2 | 1 | 1 | 1 | 4 | 5 | 3 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 9
  Not Hispanic or Latino | 3 | 7 | 0 | 5 | 2 | 3 | 4 | 3 | 1 | 3 | 2 | 7 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Asian | 0 | 7 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 0 | 3 | 4 | 1 | 0 | 3 | 1 | 1 | 4 | 2 | 6 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Permanent Discontinuation of IMP
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant administered a medicinal product which did not necessarily have a causal relationship with the IMP. TEAEs were defined as AEs which started, or worsened, after the first dose of IMP. An SAE was any untoward medical occurrence or effect that, at any dose, resulted in death; was life threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity or other important medical event.
Time Frame: From start of IMP on Day 1 up to Day 7
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants
  TEAEs | 2 | 5 | 3 | 1
  SAEs | 0 | 1 | 0 | 0
  TEAEs leading to permanent discontinuation of IMP | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Permanent Discontinuation of IMP
Description: An AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal product which did not necessarily have a causal relationship with the IMP. TEAEs were defined as AEs which started, or worsened, after the first dose of IMP. An SAE was any untoward medical occurrence or effect that, at any dose, resulted in death; was life threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity or other important medical event.
Time Frame: From start of IMP on Day 1 up to Day 12
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8
Participants
  TEAEs | 1 | 2 | 1 | 1 | 1 | 2 | 3 | 1
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to permanent discontinuation of IMP | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Physical Examination Results at Baseline
Description: Physical examination included general appearance; head, eyes, ears, nose and throat (HEENT); dermatologic, cardiovascular, respiratory, gastrointestinal and neurological examination. Clinical significance of results were determined by the investigator.
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants
  General appearance: number analyzed (Participants) | 3 | 7 | 3 | 5
  General appearance | 0 | 1 | 0 | 0
  HEENT: number analyzed (Participants) | 3 | 7 | 3 | 4
  HEENT | 1 | 2 | 0 | 0
  Dermatologic: number analyzed (Participants) | 3 | 7 | 3 | 4
  Dermatologic | 0 | 0 | 0 | 0
  Cardiovascular: number analyzed (Participants) | 3 | 7 | 3 | 5
  Cardiovascular | 0 | 1 | 0 | 0
  Respiratory: number analyzed (Participants) | 3 | 7 | 3 | 5
  Respiratory | 3 | 6 | 2 | 1
  Gastrointestinal: number analyzed (Participants) | 3 | 7 | 3 | 5
  Gastrointestinal | 0 | 0 | 0 | 0
  Neurological: number analyzed (Participants) | 3 | 7 | 3 | 5
  Neurological | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Physical Examination Results Anytime Between 18 to 24 Hours Post-dose
Description: Physical examination included general appearance, HEENT, dermatologic, cardiovascular, respiratory, gastrointestinal and neurological examination. Clinical significance of results were determined by the investigator.
Time Frame: Anytime between 18 to 24 hours post-dose on Day 1
Population: Safety population included all participants who received at least 1 dose of IMP. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants
  General appearance | 0 | 0 | 0 | 0
  HEENT: number analyzed (Participants) | 3 | 6 | 1 | 5
  HEENT | 1 | 2 | 0 | 0
  Dermatologic: number analyzed (Participants) | 3 | 6 | 1 | 5
  Dermatologic | 0 | 0 | 0 | 0
  Cardiovascular | 0 | 0 | 0 | 0
  Respiratory | 1 | 4 | 1 | 1
  Gastrointestinal | 0 | 0 | 0 | 0
  Neurological | 0 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Physical Examination Results at 48 Hours Post-dose
Description: as for outcome 4
Time Frame: At 48 hours post-dose on Day 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants
  General appearance | 0 | 0 | 0 | 0
  HEENT: number analyzed (Participants) | 3 | 6 | 2 | 5
  HEENT | 1 | 1 | 1 | 0
  Dermatologic: number analyzed (Participants) | 3 | 6 | 2 | 5
  Dermatologic | 0 | 0 | 0 | 0
  Cardiovascular | 0 | 0 | 0 | 0
  Respiratory | 1 | 3 | 1 | 1
  Gastrointestinal | 0 | 0 | 0 | 0
  Neurological | 0 | 0 | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Physical Examination Results at Baseline
Description: as for outcome 4
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 3 | 1 | 4 | 5 | 7
Participants
  General Appearance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  HEENT: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1 | 4 | 5 | 7
  HEENT | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Dermatologic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Respiratory | 1 | 2 | 3 | 3 | 1 | 2 | 4 | 3
  Gastrointestinal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neurological | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Physical Examination Results Anytime Between 40 to 48 Hours Post-dose 10
Description: as for outcome 4
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
Participants
  General appearance | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  HEENT: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 8
  HEENT | 0 | 0 | 1 | 0 |  | 0 | 0 | 0
  Dermatologic: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 8
  Dermatologic | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Cardiovascular: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 8
  Cardiovascular | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Respiratory | 0 | 1 | 0 | 0 |  | 1 | 0 | 0
  Gastrointestinal: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 8
  Gastrointestinal | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Neurological: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 8
  Neurological | 0 | 0 | 0 | 0 |  | 0 | 0 | 0

8. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Baseline
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure.
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants | 0 | 2 | 0 | 0

9. Secondary Outcome: Part A: Time to Maximum Plasma Concentration (Tmax)
Description: No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the Pharmacokinetic (PK) population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included all participants who received IMP and had at least 1 post-dose PK concentration measurement.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Hours | 4.17 (4) [4 to 4.5] | 4.58 (4.42) [4.42 to 6.18] | 7 (4.87) [4.87 to 48.3] | 4.78 (2) [2 to 6.67]

10. Secondary Outcome: Part B: Time to Maximum Plasma Concentration (Tmax)
Description: No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: Day 1 Dose 1 (anytime between 4 to 5 hours post-dose, 12 hours post-dose), Day 3 Dose 6 (pre-dose, anytime between 4 to 5 hours post-dose, 12 hours post-dose)
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 8
Hours
  Dose 1 | 4.6 [4.33 to 4.63] | 4.32 [3.58 to 11.6] | 4.17 [2.5 to 4.17] | 4.03 [3.77 to 5.5] | 4.31 [4.08 to 12]
  Dose 6: number analyzed (Participants) | 3 | 3 | 2 | 3 | 8
  Dose 6 | 4.43 [4.38 to 4.5] | 3.95 [3.67 to 4.88] | 4.53 [4.05 to 5] | 4.58 [3.58 to 11.5] | 4.29 [0 to 11.8]

11. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax)
Description: No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Nanograms per milliliter | 1.59 (2.76) [lower limit 2.76] | 8.08 (7.94) [lower limit 7.94] | 2.98 (3.09) [lower limit 3.09] | 28 (17.5) [lower limit 17.5]

12. Secondary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 8
Nanograms per milliliter
  Dose 1 | 43.2 (36.7) | 24.9 (20) | 115 (182) | 39.3 (26.4) | 56.5 (88.1)
  Dose 6: number analyzed (Participants) | 3 | 3 | 2 | 3 | 8
  Dose 6 | 30.9 (31.3) | 67.8 (86.3) | 212 (157) | 133 (64.8) | 177 (151)

13. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to 12 Hours (AUC0-12)
Description: AUC(0 to 12) was calculated using the linear trapezoidal method. No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 2 | 6
Hours*nanogram per milliliter | 9.22 (16) [lower limit 16] | 45 (48) [lower limit 48] | 6.46 (9.14) [lower limit 9.14] | 201 (143) [lower limit 143]

14. Secondary Outcome: Part B: Area Under the Plasma Concentration Time Curve From Time Zero to 12 Hours (AUC0-12)
Description: AUC(0 to 12) was calculated using the linear trapezoidal method. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4
Hours*nanogram per milliliter
  Dose 1: number analyzed (Participants) | 0 | 0 | 2 | 1 | 4
  Dose 1 |  |  | 1170 (1460) | 127 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 160 (120)
  Dose 6: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Dose 6 | 87.9 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 184 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 1110 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1600 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.

15. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUC[0 to t])
Description: Area under the plasma concentration-time curve from time 0 to the last measurable concentration was determined using the linear trapezoidal method. No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 1 | 6 | 2 | 6
Hours*nanogram per milliliter | 23.1 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 48.1 (49.9) | 14 (1.46) | 287 (217)

16. Secondary Outcome: Part B: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUC[0 to t])
Description: Area under the plasma concentration-time curve from time 0 to the last measurable concentration was determined using the linear trapezoidal method. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 4 | 2 | 4 | 8
Hours*nanogram per milliliter
  Dose 1 | 288 (251) | 163 (132) | 1170 (1460) | 342 (240) | 315 (386)
  Dose 6: number analyzed (Participants) | 3 | 3 | 2 | 3 | 8
  Dose 6 | 225 (233) | 477 (594) | 1560 (1010) | 1310 (802) | 1140 (845)

17. Secondary Outcome: Part A: Terminal Half-life (t1/2)
Description: T1/2 was calculated as loge (2) divided by kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed for Cohort 1 due to insufficient number of quantifiable sisunatovir concentrations.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 5
Hours |  |  |  | 6.22 (1.46) [lower limit 1.46]

18. Secondary Outcome: Part B: Terminal Half-life (t1/2)
Description: as for outcome 17
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed as at least 3 quantifiable concentrations were required to calculate t1/2 and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0 to Inf)
Description: AUCinf was determined as AUC(0 to t) + (Clast/kel), where Clast was the plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis and kel was the terminal phase rate. No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed for Cohort 1 as at least 3 quantifiable concentrations were required to calculate AUC(0 to inf) and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 5
Hours*nanogram per milliliter |  |  |  | 231 (161) [lower limit 161]

20. Secondary Outcome: Part B: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0 to Inf)
Description: AUCinf was determined as AUC(0 to t) + (Clast/kel), where Clast was the plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis and kel was the terminal phase rate. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed as at least 3 quantifiable concentrations were required to calculate AUC(0 to inf) and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Part A: Trough Concentration at the End of First Dosing Interval (C12)
Time Frame: At 12 hours post-dose on Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 1 | 6
Nanogram per milliliter | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | 0.851 (1.52) | 1.06 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 10.4 (9.57)

22. Secondary Outcome: Part B: Trough Concentration at the End of Dose 6 (C12)
Time Frame: At 12 hours post-dose 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 8
Nanograms per milliliter | 7.6 (8.33) [lower limit 8.33] | 9.55 (9.75) [lower limit 9.75] | 36.9 (5.3) [lower limit 5.3] | 89.8 (99.1) [lower limit 99.1] | 124 (167) [lower limit 167]

23. Secondary Outcome: Part A: Predicted Plasma Clearance
Description: Clearance was calculated as Dose divided by AUC(0 to inf). No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed for Cohort 1 as at least 3 quantifiable concentrations were required to calculate clearance and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Measure: Mean (Standard Deviation); unit: Liters per hour per kilogram
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 5
Liters per hour per kilogram |  |  |  | 12.7 (7.66) [lower limit 7.66]

24. Secondary Outcome: Part B: Predicted Plasma Clearance
Description: Clearance was calculated as Dose divided by AUC(0 to inf). No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed as at least 3 quantifiable concentrations were required to calculate clearance and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Part A: Apparent Volume of Distribution of the Drug After Extravascular Administration
Description: Apparent volume of distribution was estimated as Dose/Kel*AUC(0 to inf), where Kel=apparent first-order terminal elimination rate constant. No sampling was done at pre-dose (0 hour) and pre-dose results were imputed for all participants in the PK population.
Time Frame: Anytime between 4 to 5 hours, anytime between 6 to 8 hours, 12 hours, 18 to 24 hours and 48 hours post-dose on Day 1
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed for Cohort 1 as at least 3 quantifiable concentrations were required to calculate volume of distribution and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Measure: Mean (Standard Deviation); unit: Litres per kilogram
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 5
Litres per kilogram |  |  |  | 119 (87.4) [lower limit 87.4]

26. Secondary Outcome: Part B: Apparent Volume of Distribution of the Drug After Extravascular Administration
Description: Apparent volume of distribution was estimated as Dose/Kel*AUC(0 to inf), where Kel=apparent first-order terminal elimination rate constant. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Analysis could not be performed as at least 3 quantifiable concentrations were required to calculate volume of distribution and this criteria could not be fulfilled due to insufficient number of quantifiable concentrations.
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Part B: Accumulation Ratio
Description: Accumulation ratio was calculated as ratio of the area under the curve (AUC) during a single dosing interval under steady state conditions to the AUC during a dosing interval after one singe dose. No sampling was done at pre-dose (0 hour) on Day 1 and pre-dose results were imputed for all participants in the PK population.
Time Frame: as for outcome 10
Population: PK population included all participants who received IMP and had at least 1 post-dose PK concentration measurement. Here, 'Overall Number of Participants Analyzed' signifies participants with evaluable data for this PK parameter. Accumulation ratio could not be calculated as it was depended on AUC which was not calculable due to insufficient number of quantifiable concentrations.
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Part B: Percentage Fluctuation
Description: Percentage fluctuation was calculated as 100*(Cmax-Cmin)/Cavg, where Cmin=minimum plasma concentration and Cmax measured over dosing interval.
Time Frame: Day 3 Dose 6 (pre-dose, anytime between 4 to 5 hours post-dose, 12 hours post-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of fluctuation
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
Percentage of fluctuation | 132 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 123 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 8.63 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 98.1 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.

29. Secondary Outcome: Part B: Area Under the Plasma Concentration Time Curve From Time Zero to the End of Last Dosing Interval (AUC0-tau)
Description: AUC(0 to tau) was determined using the linear trapezoidal method.
Time Frame: Day 3 Dose 6 (pre-dose, anytime between 4 to 5 hours post-dose, 12 hours post-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
Hours*nanogram per milliliter | 87.9 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 184 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 1110 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1600 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.

30. Secondary Outcome: Part B: Average Plasma Concentration Over Dosing Interval (Cavg)
Description: Cavg was estimated as AUC(0 to tau)/tau, where tau=dosing interval (12 hours).
Time Frame: Day 3 Dose 6 (pre-dose, anytime between 4 to 5 hours post-dose, 12 hours post-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
Nanogram per milliliter | 7.32 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 15.3 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 92.7 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 133 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.

31. Secondary Outcome: Part B: Minimum Observed Plasma Concentration
Time Frame: Day 3 Dose 6 (pre-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 8
Nanograms per milliliter | 8.51 (9.87) | 24.3 (24.7) | 70.8 (20.9) | 96.7 (48.6) | 59.6 (65.7)

32. Secondary Outcome: Part B: Plasma Trough Concentration
Time Frame: Day 3 Dose 6 (pre-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: RV521 2.5 mg/kg | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 8
Nanograms per milliliter | 8.51 (9.87) | 24.3 (24.7) | 70.8 (20.9) | 96.7 (48.6) | 59.6 (65.7)

33. Secondary Outcome: Part B: Percent Change From Baseline in Logarithm to Base10 (Log10) Total RSV Viral Load by Quantitative Reverse Transcription Polymerase Chain Reaction (RT-qPCR)
Description: Percent change from baseline in log10 total RSV viral load was analyzed using a mixed effects analysis of covariance (ANCOVA) model. The model was fitted to the participants treated at the final doses selected for Cohort 5 as pre-planned in statistical analysis plan for age group >=1 month to <6 months.
Time Frame: Baseline (pre-dose on Day 1), 60 hours and 156 hours after first dose on Day 1
Population: Modified Intent to Treat (mITT) population included all participants who received at least 1 dose of IMP (RV521 or placebo) and had a pre-treatment positive RSV nasopharyngeal swab confirmed by the central laboratory and agreed by the project team during blind data review meeting. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoints. Data for Cohorts 4 and 5 were combined as pre-specified in statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Cohort 4 and 5 Combined: Placebo: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received BID of placebo separated by 12 hours orally for 5 days. Participants from Cohorts 4 and 5 were included.
- Cohort 4 and 5 Combined: RV521 2.5 mg/kg: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received BID of RV521 2.5 mg/kg separated by 12 hours orally for 5 days. Participants from Cohort 4 and 5 were included.
Arm/Group | Cohort 4 and 5 Combined: Placebo | Cohort 4 and 5 Combined: RV521 2.5 mg/kg
Number analyzed (Participants) | 6 | 12
Percent change
  60 hours: number analyzed (Participants) | 5 | 11
  60 hours | -23.27 (10.48) | -31.29 (8.19)
  156 hours: number analyzed (Participants) | 4 | 12
  156 hours | -32.31 (11.52) | -47.53 (8.03)
Statistical Analysis 1: Comparison: Cohort 4 and 5 Combined: Placebo vs Cohort 4 and 5 Combined: RV521 2.5 mg/kg; 60 hours. Analysis was performed using mixed effects analysis of covariance model on change from baseline in viral load, including a random effect for participant and fixed effects for treatment group, baseline human rhinovirus/enterovirus status (present or absent), visit, vist by treatment group interaction, and baseline viral load as a covariate; Test type: Other; Difference = -8.02, 95% CI 2-sided [-31.78 to 15.74]
Statistical Analysis 2: Comparison: Cohort 4 and 5 Combined: Placebo vs Cohort 4 and 5 Combined: RV521 2.5 mg/kg; 156 hours. Analysis was performed using mixed effects analysis of covariance model on change from baseline in viral load, including a random effect for participant and fixed effects for treatment group, baseline human rhinovirus/enterovirus status (present or absent), visit, vist by treatment group interaction, and baseline viral load as a covariate; Test type: Other; Mixed effects analysis of covariance; Difference = -15.22, 95% CI 2-sided [-40.15 to 9.70]

34. Secondary Outcome: Part B: Percent Change From Baseline in Logarithm to Base10 (Log10) Total RSV Viral Load by Cell-Based Infectivity Assay (CBIA)
Description: Percent change from baseline in log10 total RSV viral load was analyzed using a mixed effects ANCOVA model. The model was fitted to the participants treated at the final doses selected for Cohort 5 as pre-planned in statistical analysis plan for age group >=1 month to <6 months.
Time Frame: Baseline (pre-dose on Day 1), 60 hours and 156 hours after first dose on Day 1
Population: mITT population included all participants who received at least 1 dose of IMP (RV521 or placebo) and had a pre-treatment positive RSV nasopharyngeal swab confirmed by the central laboratory and agreed by the project team during blind data review meeting. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoints. Data for Cohorts 4 and 5 were combined as pre-specified in statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 4 and 5 Combined: Placebo | Cohort 4 and 5 Combined: RV521 2.5 mg/kg
Number analyzed (Participants) | 6 | 12
Percent change
  60 hours: number analyzed (Participants) | 5 | 11
  60 hours | -69.56 (46.32) | -54.74 (34.87)
  156 hours: number analyzed (Participants) | 4 | 12
  156 hours | -10.00 (51.88) | -41.20 (34.01)
Statistical Analysis 1: Comparison: Cohort 4 and 5 Combined: Placebo vs Cohort 4 and 5 Combined: RV521 2.5 mg/kg; [analysis description as in outcome 33, analysis 1]; Test type: Other; Difference = 14.82, 95% CI 2-sided [-91.68 to 121.33]
Statistical Analysis 2: Comparison: Cohort 4 and 5 Combined: Placebo vs Cohort 4 and 5 Combined: RV521 2.5 mg/kg; [analysis description as in outcome 33, analysis 2]; Test type: Other; Difference = -31.19, 95% CI 2-sided [-143.96 to 81.57]

35. Secondary Outcome: Part B: Time to Resolution of RSV-Related Signs and Symptoms
Description: Time to resolution was calculated for RSV-related signs and symptoms that were present at study start and was defined as the time of randomization to the time that RSV-related signs and symptoms were absent.
Time Frame: Up to Day 12
Population: mITT population included all participants who received at least 1 dose of IMP (RV521 or placebo) and had a pre-treatment positive RSV nasopharyngeal swab confirmed by the central laboratory and agreed by the project team during blind data review meeting. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Days | 6.20 (6.1) [6.1 to 6.6] | 6.20 (6.2) [6.2 to 6.3] | 6.45 (5.9) [5.9 to 6.8] | 3.80 (2.6) [2.6 to 5.0] | 4.90 (4.9) [4.9 to 4.9] | 6.30 (4.6) [4.6 to 6.9] | 6.00 (2.5) [2.5 to 6.7] | 6.10 (4.1) [4.1 to 6.9]

36. Secondary Outcome: Part B: Time to Improvement in RSV-Related Signs and Symptoms
Description: Time to improvement was calculated for RSV-related signs and symptoms that were classified as moderate or severe during the course of the study and was defined as the time from randomization to the time that RSV-related signs and symptoms were mild or absent.
Time Frame: Up to Day 12
Population: as for outcome 35
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Days | 2.25 (1.5) [1.5 to 3.0] | 0.50 (0.5) [0.5 to 6.3] | 3.15 (2.1) [2.1 to 5.9] | 2.55 (1.1) [1.1 to 4.0] | 1.90 (1.9) [1.9 to 1.9] | 4.35 (3.6) [3.6 to 6.9] | 3.00 (1.0) [1.0 to 6.0] | 6.00 (1.5) [1.5 to 6.9]

37. Secondary Outcome: Part B: RSV Clinical Scoring System Scores
Description: RSV clinical score was a composite score for infants with RSV infection >= 1 month of age based on 4 items (respiratory rate, wheezing, retraction of respiratory muscles and general condition). Score for each item ranged from 0 to 3 where 0=none/normal and 3=severe. Total score was calculated as sum of individual items and ranged from 0 to 12, where higher score indicated severe disease. RSV symptoms were graded as mild: score <=5, moderate: score > 5 but < 9 and severe: score >=9.
Time Frame: Baseline (pre-dose 1 on Day 1), pre-dose 3, pre-dose 5, pre-dose 7, pre-dose 9, anytime between 40 to 48 hours post-dose 10 on Day 5
Population: mITT population included all participants who received at least 1 dose of IMP (RV521 or placebo) and had a pre-treatment positive RSV nasopharyngeal swab confirmed by the central laboratory and agreed by the project team during blind data review meeting. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Units on a scale
  Baseline: number analyzed (Participants) | 2 | 3 | 4 | 2 | 1 | 4 | 5 | 8
  Baseline | 3.5 (2.12) | 5.0 (1.73) | 6.8 (2.50) | 4.5 (6.36) | 8.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 6.8 (2.22) | 6.2 (3.56) | 6.0 (2.73)
  pre-dose 3 | 2.0 (1.73) | 4.0 (2.65) | 2.5 (1.29) | 1.0 (1.41) | 4.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 5.0 (0.00) | 1.8 (1.10) | 4.3 (2.38)
  pre-dose 5 | 1.0 (1.00) | 2.7 (2.08) | 1.8 (1.50) | 2.5 (3.54) | 3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.3 (0.96) | 1.4 (1.14) | 3.9 (2.75)
  pre-dose 7: number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 3 | 5 | 8
  pre-dose 7 | 0.7 (0.58) | 3.0 (1.73) | 1.3 (1.50) | 2.5 (3.54) | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1.3 (0.58) | 1.6 (0.55) | 2.3 (2.12)
  pre-dose 9: number analyzed (Participants) | 1 | 2 | 2 | 1 | 1 | 2 | 4 | 4
  pre-dose 9 | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (2.12) | 1.5 (0.71) | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 2.0 (1.41) | 1.8 (0.50) | 2.3 (0.96)
  40 to 48 hours post-dose 10: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 3 | 5 | 8
  40 to 48 hours post-dose 10 | 0.3 (0.58) | 1.0 (1.00) | 0.5 (0.58) | 0.0 (0.00) |  | 1.0 (1.00) | 1.2 (1.10) | 0.6 (0.52)

38. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose
Description: as for outcome 8
Time Frame: Anytime between 4 to 5 hours post-dose on Day 1
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants | 0 | 1 | 1 | 0

39. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at 12 Hours Post-Dose
Description: as for outcome 8
Time Frame: At 12 hours post-dose on Day 1
Population: Safety population included all participants who received at least 1 dose of IMP. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 2 | 6
Participants | 0 | 2 | 0 | 0

40. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation Anytime Between 18 to 24 Hours Post-Dose
Description: as for outcome 8
Time Frame: Anytime between 18 to 24 hours post-dose on Day 1
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants | 0 | 2 | 0 | 0

41. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at 48 Hours Post-Dose
Description: as for outcome 8
Time Frame: 48 hours post-dose on Day 1
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants | 0 | 1 | 0 | 0

42. Primary Outcome: Part B: Number of Participants With Abnormal Vital Signs Per Investigator's Interpretation at Baseline
Description: as for outcome 8
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose 1
Description: as for outcome 8
Time Frame: Anytime between 4 to 5 hours post-dose 1 (Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation At Pre-dose 2
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 2= assessment prior to receiving dose 2 of IMP on Day 1.
Time Frame: Pre-dose 2 (Day 1)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

45. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 3
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 3= assessment prior to receiving dose 3 of IMP on Day 2.
Time Frame: Pre-dose 3 (Day 2)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 4
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 4= assessment prior to receiving dose 4 of IMP on Day 2.
Time Frame: Pre-dose 4 (Day 2)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

47. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 5
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 5= assessment prior to receiving dose 5 of IMP on Day 3.
Time Frame: Pre-dose 5 (Day 3)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

48. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 6
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 6= assessment prior to receiving dose 6 of IMP on Day 3.
Time Frame: Pre-dose 6 (Day 3)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 3 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose 6
Description: as for outcome 8
Time Frame: Anytime between 4 to 5 hours post-dose 6 (Day 3)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 7
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 7= assessment prior to receiving dose 7 of IMP on Day 4.
Time Frame: Pre-dose 7 (Day 4)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 3 | 5 | 8
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

51. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 8
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 8= assessment prior to receiving dose 8 of IMP on Day 4.
Time Frame: Pre-dose 8 (Day 4)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 3 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

52. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 9
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 9= assessment prior to receiving dose 9 of IMP on Day 5.
Time Frame: Pre-dose 9 (Day 5)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 2 | 2 | 1 | 1 | 3 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

53. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation at Pre-dose 10
Description: Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate, heart rate and pulse oximetry. Number of participants with abnormal clinically significant vital signs per investigator's interpretation are reported in this outcome measure. Predose 10= assessment prior to receiving dose 10 of IMP on Day 5.
Time Frame: Pre-dose 10 (Day 5)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 1 | 3 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

54. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Vital Signs Per Investigator's Interpretation Anytime Between 40 to 48 Hours Post-Dose 10
Description: as for outcome 8
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 |  | 0 | 0 | 0

55. Primary Outcome: Part A: Number of Participants With Abnormal Hematology Results at Baseline
Description: Hematology parameters included basophils, eosinophils, mean cell hemoglobin concentration (MCHC), mean cell hemoglobin (MCH), mean cell volume (MCV), red blood cell count (RBC), hematocrit (HCT), hemoglobin (Hb), white blood cell count (WBC), lymphocytes, monocytes, neutrophils and platelet count. Institutional laboratory normal ranges were used.
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 2 | 7 | 3 | 6
Participants
  Basophils; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Basophils; below normal range | 0 | 0 | 0 | 0
  Basophils; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Basophils; above normal range | 0 | 0 | 0 | 0
  Eosinophils; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Eosinophils; below normal range | 0 | 0 | 0 | 0
  Eosinophils; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Eosinophils; above normal range | 0 | 0 | 0 | 0
  MCHC; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCHC; below normal range | 0 | 0 | 0 | 0
  MCHC; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCHC; above normal range | 0 | 0 | 0 | 0
  MCH; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCH; below normal range | 0 | 0 | 0 | 0
  MCH; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCH; above normal range | 0 | 0 | 0 | 0
  MCV; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCV; below normal range | 0 | 0 | 0 | 0
  MCV; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  MCV; above normal range | 0 | 0 | 0 | 0
  RBC; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  RBC; below normal range | 0 | 0 | 0 | 0
  RBC; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  RBC; above normal range | 0 | 0 | 0 | 0
  HCT; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  HCT; below normal range | 0 | 0 | 0 | 0
  HCT; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  HCT; above normal range | 0 | 0 | 0 | 0
  Hb; below normal range | 0 | 0 | 1 | 0
  Hb; above normal range | 0 | 0 | 0 | 0
  WBC; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  WBC; below normal range | 0 | 0 | 1 | 1
  WBC; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  WBC; above normal range | 0 | 0 | 0 | 0
  Lymphocytes; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Lymphocytes; below normal range | 0 | 0 | 0 | 0
  Lymphocytes; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Lymphocytes; above normal range | 0 | 0 | 0 | 0
  Monocytes; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Monocytes; below normal range | 0 | 0 | 0 | 0
  Monocytes; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Monocytes; above normal range | 0 | 0 | 0 | 0
  Neutrophils; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Neutrophils; below normal range | 0 | 0 | 0 | 0
  Neutrophils; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Neutrophils; above normal range | 0 | 0 | 0 | 0
  Platelets; below normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Platelets; below normal range | 0 | 2 | 0 | 1
  Platelets; above normal range: number analyzed (Participants) | 2 | 7 | 1 | 6
  Platelets; above normal range | 0 | 0 | 0 | 1

56. Primary Outcome: Part A: Number of Participants With Abnormal Hematology Results at 48 Hours Post-Dose
Description: Hematology parameters included basophils, eosinophils, MCHC, MCH, MCV, RBC, HCT, Hb, WBC, lymphocytes, monocytes, neutrophils and platelet count. Institutional laboratory normal ranges were used.
Time Frame: At 48 hours post-dose on Day 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 5
Participants
  Basophils; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Basophils; below normal range | 0 | 0 | 0 | 0
  Basophils; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Basophils; above normal range | 0 | 0 | 0 | 0
  Eosinophils; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Eosinophils; below normal range | 0 | 0 | 0 | 0
  Eosinophils; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Eosinophils; above normal range | 0 | 0 | 0 | 0
  MCHC; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCHC; below normal range | 0 | 0 | 0 | 0
  MCHC; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCHC; above normal range | 0 | 0 | 0 | 0
  MCH; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCH; below normal range | 0 | 0 | 0 | 0
  MCH; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCH; above normal range | 0 | 0 | 0 | 0
  MCV; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCV; below normal range | 0 | 0 | 0 | 0
  MCV; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  MCV; above normal range | 0 | 0 | 0 | 0
  RBC; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  RBC; below normal range | 0 | 0 | 0 | 0
  RBC; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  RBC; above normal range | 0 | 0 | 0 | 0
  HCT; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  HCT; below normal range | 0 | 0 | 0 | 0
  HCT; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  HCT; above normal range | 0 | 0 | 0 | 0
  Hb; below normal range | 0 | 0 | 0 | 0
  Hb; above normal range | 0 | 0 | 0 | 0
  WBC; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  WBC; below normal range | 0 | 0 | 0 | 0
  WBC; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  WBC; above normal range | 0 | 0 | 0 | 1
  Lymphocytes; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Lymphocytes; below normal range | 0 | 0 | 0 | 0
  Lymphocytes; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Lymphocytes; above normal range | 0 | 0 | 0 | 0
  Monocytes; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Monocytes; below normal range | 0 | 0 | 0 | 0
  Monocytes; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Monocytes; above normal range | 0 | 0 | 0 | 0
  Neutrophils; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Neutrophils; below normal range | 0 | 0 | 0 | 0
  Neutrophils; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Neutrophils; above normal range | 0 | 0 | 0 | 0
  Platelets; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Platelets; below normal range | 0 | 1 | 0 | 0
  Platelets; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Platelets; above normal range | 1 | 1 | 1 | 1

57. Primary Outcome: Part B: Number of Participants With Abnormal Hematology Results at Baseline
Description: as for outcome 56
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 0 | 4 | 2 | 7
Participants
  Basophils; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Basophils; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Eosinophils; below normal range | 1 | 0 | 1 | 0 |  | 0 | 0 | 2
  Eosinophils; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  MCHC; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  MCHC; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  MCH; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  MCH; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  MCV; below normal range | 0 | 0 | 1 | 0 |  | 0 | 0 | 0
  MCV; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  RBC; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  RBC; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  HCT; below normal range | 0 | 0 | 0 | 1 |  | 0 | 2 | 0
  HCT; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Hb; below normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 1
  Hb; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  WBC; below normal range | 0 | 0 | 0 | 0 |  | 2 | 1 | 0
  WBC; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Lymphocytes; below normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 0
  Lymphocytes; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Monocytes; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Monocytes; above normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  Neutrophils; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Neutrophils; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Platelets; below normal range: number analyzed (Participants) | 3 | 3 | 3 | 1 | 0 | 3 | 2 | 7
  Platelets; below normal range | 1 | 0 | 1 | 0 |  | 0 | 0 | 0
  Platelets; above normal range: number analyzed (Participants) | 3 | 3 | 3 | 1 | 0 | 3 | 2 | 7
  Platelets; above normal range | 1 | 0 | 0 | 0 |  | 0 | 0 | 1

58. Primary Outcome: Part B: Number of Participants With Abnormal Hematology Results Anytime Between 40 to 48 Hours Post-dose 10
Description: as for outcome 56
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 2 | 4 | 2 | 0 | 1 | 3 | 7
Participants
  Basophils; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Basophils; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Eosinophils; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Eosinophils; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  MCHC; below normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 1
  MCHC; above normal range | 0 | 0 | 0 | 1 |  | 0 | 0 | 0
  MCH; below normal range | 0 | 0 | 0 | 1 |  | 0 | 0 | 1
  MCH; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  MCV; below normal range | 0 | 0 | 1 | 1 |  | 0 | 0 | 0
  MCV; above normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 0
  RBC; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  RBC; above normal range | 0 | 0 | 2 | 1 |  | 0 | 1 | 0
  HCT; below normal range | 0 | 0 | 0 | 0 |  | 0 | 2 | 0
  HCT; above normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 0
  Hb; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Hb; above normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 0
  WBC; below normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  WBC; above normal range | 1 | 0 | 0 | 0 |  | 0 | 0 | 0
  Lymphocytes; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Lymphocytes; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Monocytes; below normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 1
  Monocytes; above normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 1
  Neutrophils; below normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  Neutrophils; above normal range | 0 | 0 | 1 | 0 |  | 0 | 1 | 0
  Platelets; below normal range: number analyzed (Participants) | 3 | 2 | 3 | 1 | 0 | 1 | 3 | 7
  Platelets; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Platelets; above normal range: number analyzed (Participants) | 3 | 2 | 3 | 1 | 0 | 1 | 3 | 7
  Platelets; above normal range | 2 | 1 | 2 | 0 |  | 0 | 2 | 6

59. Primary Outcome: Part A: Number of Participants With Abnormal Clinical Chemistry Results at Baseline
Description: Clinical chemistry parameters included alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin, calcium, chloride, creatinine, gamma glutamyltransferase (GGT), glucose, lactate dehydrogenase (LDH), potassium, protein, sodium and urea. Institutional laboratory normal ranges were used.
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants
  ALT; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  ALT; below normal range | 0 | 0 | 0 | 0
  ALT; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  ALT; above normal range | 0 | 0 | 0 | 0
  Albumin; below normal range | 0 | 0 | 0 | 0
  Albumin; above normal range | 0 | 0 | 0 | 0
  ALP; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  ALP; below normal range | 0 | 0 | 0 | 0
  ALP; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  ALP; above normal range | 0 | 0 | 0 | 0
  AST; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  AST; below normal range | 0 | 0 | 0 | 0
  AST; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  AST; above normal range | 0 | 0 | 0 | 0
  Bilirubin; below normal range | 0 | 0 | 0 | 0
  Bilirubin; above normal range | 0 | 0 | 0 | 0
  Calcium; below normal range | 0 | 1 | 0 | 0
  Calcium; above normal range | 0 | 0 | 0 | 1
  Chloride; below normal range | 0 | 0 | 0 | 0
  Chloride; above normal range | 0 | 0 | 0 | 0
  Creatinine; below normal range | 0 | 0 | 0 | 0
  Creatinine; above normal range | 0 | 0 | 0 | 0
  GGT; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  GGT; below normal range | 0 | 0 | 0 | 0
  GGT; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 5
  GGT; above normal range | 0 | 0 | 0 | 0
  Glucose; below normal range | 0 | 0 | 0 | 0
  Glucose; above normal range | 0 | 0 | 0 | 0
  LDH; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 3
  LDH; below normal range | 0 | 0 | 0 | 0
  LDH; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 3
  LDH; above normal range | 0 | 0 | 0 | 0
  Potassium; below normal range: number analyzed (Participants) | 3 | 7 | 3 | 4
  Potassium; below normal range | 0 | 0 | 0 | 0
  Potassium; above normal range: number analyzed (Participants) | 3 | 7 | 3 | 4
  Potassium; above normal range | 0 | 0 | 0 | 1
  Protein; below normal range | 0 | 0 | 0 | 0
  Protein; above normal range | 0 | 0 | 0 | 0
  Sodium; below normal range | 0 | 1 | 0 | 0
  Sodium; above normal range | 0 | 0 | 0 | 0
  Urea; below normal range | 0 | 0 | 0 | 0
  Urea; above normal range | 0 | 0 | 0 | 0

60. Primary Outcome: Part A: Number of Participants With Abnormal Clinical Chemistry Results at 48 Hours Post-Dose
Description: Clinical chemistry parameters included ALT, albumin, ALP, AST, bilirubin, calcium, chloride, creatinine, GGT, glucose, LDH, potassium, protein, sodium and urea. Institutional laboratory normal ranges were used.
Time Frame: At 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 1 | 6
Participants
  ALT; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  ALT; below normal range | 0 | 0 | 0 | 0
  ALT; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  ALT; above normal range | 0 | 0 | 0 | 0
  Albumin; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Albumin; below normal range | 0 | 0 | 0 | 0
  Albumin; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Albumin; above normal range | 0 | 0 | 0 | 0
  ALP; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  ALP; below normal range | 0 | 0 | 0 | 0
  ALP; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  ALP; above normal range | 0 | 0 | 0 | 0
  AST; below normal range: number analyzed (Participants) | 3 | 5 | 1 | 5
  AST; below normal range | 0 | 0 | 0 | 0
  AST; above normal range: number analyzed (Participants) | 3 | 5 | 1 | 5
  AST; above normal range | 0 | 0 | 0 | 0
  Bilirubin; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Bilirubin; below normal range | 0 | 0 | 0 | 0
  Bilirubin; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Bilirubin; above normal range | 0 | 0 | 0 | 0
  Calcium; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Calcium; below normal range | 0 | 0 | 0 | 0
  Calcium; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Calcium; above normal range | 0 | 0 | 0 | 1
  Chloride; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Chloride; below normal range | 0 | 0 | 0 | 0
  Chloride; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Chloride; above normal range | 0 | 0 | 0 | 0
  Creatinine; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 4
  Creatinine; below normal range | 0 | 0 | 0 | 0
  Creatinine; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 4
  Creatinine; above normal range | 0 | 0 | 0 | 0
  GGT; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  GGT; below normal range | 0 | 0 | 0 | 0
  GGT; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  GGT; above normal range | 0 | 0 | 0 | 0
  Glucose; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 4
  Glucose; below normal range | 0 | 0 | 0 | 1
  Glucose; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 4
  Glucose; above normal range | 0 | 0 | 0 | 0
  LDH; below normal range: number analyzed (Participants) | 3 | 5 | 1 | 5
  LDH; below normal range | 0 | 0 | 0 | 0
  LDH; above normal range: number analyzed (Participants) | 3 | 5 | 1 | 5
  LDH; above normal range | 0 | 0 | 0 | 0
  Potassium; below normal range: number analyzed (Participants) | 3 | 5 | 1 | 4
  Potassium; below normal range | 0 | 0 | 0 | 0
  Potassium; above normal range: number analyzed (Participants) | 3 | 5 | 1 | 4
  Potassium; above normal range | 0 | 1 | 0 | 3
  Protein; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Protein; below normal range | 0 | 0 | 0 | 0
  Protein; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Protein; above normal range | 0 | 0 | 0 | 0
  Sodium; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Sodium; below normal range | 0 | 0 | 0 | 0
  Sodium; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Sodium; above normal range | 0 | 0 | 0 | 0
  Urea; below normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Urea; below normal range | 0 | 0 | 0 | 0
  Urea; above normal range: number analyzed (Participants) | 3 | 6 | 1 | 5
  Urea; above normal range | 0 | 0 | 0 | 0

61. Primary Outcome: Part B: Number of Participants With Abnormal Clinical Chemistry Results at Baseline
Description: as for outcome 60
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8
Participants
  ALT; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 0 | 4 | 5 | 8
  ALT; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  ALT; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 0 | 4 | 5 | 8
  ALT; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 3
  Albumin; below normal range: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1 | 4 | 4 | 8
  Albumin; below normal range | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Albumin; above normal range: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1 | 4 | 4 | 8
  Albumin; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALP; below normal range: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1 | 4 | 4 | 5
  ALP; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP; above normal range: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1 | 4 | 4 | 5
  ALP; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 0 | 4 | 5 | 7
  AST; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  AST; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 0 | 4 | 5 | 7
  AST; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Bilirubin; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  Bilirubin; below normal range | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2
  Bilirubin; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  Bilirubin; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 4 | 3 | 6
  Calcium; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Calcium; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 4 | 3 | 6
  Calcium; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Chloride; below normal range | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; below normal range | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 4
  Creatinine; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT; below normal range: number analyzed (Participants) | 2 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  GGT; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT; above normal range: number analyzed (Participants) | 2 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  GGT; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  Glucose; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 8
  Glucose; above normal range | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 4
  LDH; below normal range: number analyzed (Participants) | 0 | 3 | 2 | 3 | 0 | 2 | 2 | 3
  LDH; below normal range |  | 0 | 0 | 0 |  | 0 | 0 | 0
  LDH; above normal range: number analyzed (Participants) | 0 | 3 | 2 | 3 | 0 | 2 | 2 | 3
  LDH; above normal range |  | 0 | 0 | 1 |  | 0 | 0 | 0
  Potassium; below normal range: number analyzed (Participants) | 1 | 3 | 3 | 3 | 0 | 3 | 5 | 7
  Potassium; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Potassium; above normal range: number analyzed (Participants) | 1 | 3 | 3 | 3 | 0 | 3 | 5 | 7
  Potassium; above normal range | 0 | 1 | 0 | 1 |  | 0 | 1 | 2
  Protein; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 7
  Protein; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Protein; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 7
  Protein; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium; below normal range | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium; above normal range | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urea; below normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 1 | 4 | 5 | 8
  Urea; below normal range | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Urea; above normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 1 | 4 | 5 | 8
  Urea; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

62. Primary Outcome: Part B: Number of Participants With Abnormal Clinical Chemistry Results Anytime Between 40 to 48 Hours Post-dose 10
Description: as for outcome 60
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 0 | 4 | 5 | 8
Participants
  ALT; below normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 3 | 5 | 6
  ALT; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  ALT; above normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 3 | 5 | 6
  ALT; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Albumin; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 6
  Albumin; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Albumin; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 6
  Albumin; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  ALP; below normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 4 | 7
  ALP; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  ALP; above normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 4 | 7
  ALP; above normal range | 0 | 0 | 1 | 0 |  | 0 | 0 | 0
  AST; below normal range: number analyzed (Participants) | 3 | 3 | 2 | 2 | 0 | 2 | 4 | 7
  AST; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  AST; above normal range: number analyzed (Participants) | 3 | 3 | 2 | 2 | 0 | 2 | 4 | 7
  AST; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Bilirubin; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 6
  Bilirubin; below normal range | 1 | 0 | 1 | 0 |  | 0 | 0 | 1
  Bilirubin; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 6
  Bilirubin; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Calcium; below normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 7
  Calcium; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Calcium; above normal range: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 4 | 5 | 7
  Calcium; above normal range | 0 | 1 | 1 | 0 |  | 1 | 0 | 5
  Chloride; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Chloride; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Chloride; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Chloride; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Creatinine; below normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Creatinine; below normal range | 1 | 0 | 0 | 1 |  | 0 | 1 | 4
  Creatinine; above normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Creatinine; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  GGT; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 7
  GGT; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  GGT; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 7
  GGT; above normal range | 0 | 0 | 0 | 1 |  | 0 | 1 | 0
  Glucose; below normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Glucose; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Glucose; above normal range: number analyzed (Participants) | 2 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Glucose; above normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  LDH; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 2 | 3 | 6
  LDH; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  LDH; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 2 | 3 | 6
  LDH; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 1
  Potassium; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 0 | 2 | 4 | 6
  Potassium; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Potassium; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 0 | 2 | 4 | 6
  Potassium; above normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  Protein; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 7
  Protein; below normal range | 0 | 0 | 0 | 0 |  | 0 | 1 | 1
  Protein; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 4 | 7
  Protein; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Sodium; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Sodium; below normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Sodium; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Sodium; above normal range | 0 | 0 | 0 | 1 |  | 0 | 0 | 0
  Urea; below normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Urea; below normal range | 1 | 0 | 1 | 1 |  | 0 | 1 | 0
  Urea; above normal range: number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
  Urea; above normal range | 0 | 0 | 0 | 0 |  | 0 | 0 | 0

63. Primary Outcome: Part A: Number of Participants With Abnormal Urinalysis Results at Baseline
Description: Following urine parameters were analyzed: epithelial cells (normal range: 0 to 5 cells per high power field [hpf]), erythrocytes (0 to 2 per hpf), granular casts (0 per low power field [lpf]), hyaline casts (0 to 1 per lpf), leukocytes (0 to 5 per hpf), RBC casts (0 per lpf), WBC casts (0 per lpf), waxy casts (0 per lpf) and pH (5 to 8).
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 2 | 7 | 3 | 6
Participants
  Epithelial Cells; below normal range | 0 | 0 | 0 | 0
  Epithelial Cells; above normal range | 0 | 0 | 0 | 0
  Erythrocytes; below normal range | 0 | 0 | 0 | 0
  Erythrocytes; above normal range | 0 | 0 | 0 | 0
  Granular casts; below normal range | 0 | 0 | 0 | 0
  Granular casts; above normal range | 0 | 0 | 0 | 0
  Hyaline casts; below normal range | 0 | 0 | 0 | 0
  Hyaline casts; above normal range | 0 | 0 | 0 | 0
  Leukocytes; below normal range | 0 | 0 | 0 | 0
  Leukocytes; above normal range | 0 | 0 | 0 | 0
  RBC cast; below normal range | 0 | 0 | 0 | 0
  RBC cast; above normal range | 0 | 0 | 0 | 0
  WBC cast; below normal range | 0 | 0 | 0 | 0
  WBC cast; above normal range | 0 | 0 | 0 | 0
  Waxy cast; below normal range | 0 | 0 | 0 | 0
  Waxy cast; above normal range | 0 | 0 | 0 | 0
  pH; below normal range: number analyzed (Participants) | 2 | 7 | 3 | 4
  pH; below normal range | 0 | 0 | 0 | 0
  pH; above normal range: number analyzed (Participants) | 2 | 7 | 3 | 4
  pH; above normal range | 0 | 1 | 0 | 0

64. Primary Outcome: Part A: Number of Participants With Abnormal Urinalysis Results at 48 Hours Post-dose
Description: Following urine parameters were analyzed: epithelial cells (normal range: 0 to 5 cells per hpf), erythrocytes (0 to 2 per hpf), granular casts (0 per lpf), hyaline casts (0 to 1 per lpf), leukocytes (0 to 5 per hpf), RBC casts (0 per lpf), WBC casts (0 per lpf), waxy casts (0 per lpf) and potential of hydrogen (pH) (5 to 8).
Time Frame: At 48 hours post-dose on Day 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 0 | 6
Participants
  Epithelial Cells; below normal range | 0 | 0 |  | 0
  Epithelial Cells; above normal range | 0 | 0 |  | 0
  Erythrocytes; below normal range | 0 | 0 |  | 0
  Erythrocytes; above normal range | 1 | 0 |  | 1
  Granular casts; below normal range | 0 | 0 |  | 0
  Granular casts; above normal range | 0 | 0 |  | 0
  Hyaline casts; below normal range | 0 | 0 |  | 0
  Hyaline casts; above normal range | 0 | 0 |  | 0
  Leukocytes; below normal range | 0 | 0 |  | 0
  Leukocytes; above normal range | 0 | 0 |  | 0
  RBC cast; below normal range | 0 | 0 |  | 0
  RBC cast; above normal range | 0 | 0 |  | 0
  WBC cast; below normal range | 0 | 0 |  | 0
  WBC cast; above normal range | 0 | 0 |  | 0
  Waxy cast; below normal range | 0 | 0 |  | 0
  Waxy cast; above normal range | 0 | 0 |  | 0
  pH; below normal range: number analyzed (Participants) | 2 | 6 | 0 | 5
  pH; below normal range | 0 | 0 |  | 0
  pH; above normal range: number analyzed (Participants) | 2 | 6 | 0 | 5
  pH; above normal range | 0 | 2 |  | 1

65. Primary Outcome: Part B: Number of Participants With Abnormal Urinalysis Results at Baseline
Description: Following urine parameters were analyzed: epithelial cells (normal range: 0 to 5 cells per hpf), erythrocytes (0 to 2 per hpf), granular casts (0 per lpf), hyaline casts (0 to 1 per lpf), leukocytes (0 to 5 per hpf), RBC casts (0 per lpf), WBC casts (0 per lpf), waxy casts (0 per lpf) and pH (5 to 8).
Time Frame: Baseline (pre-dose on Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 2 | 4 | 5
Participants
  Epithelial cells; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Epithelial cells; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Epithelial cells; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Epithelial cells; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 2 | 4 | 3
  Erythrocytes; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Erythrocytes; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 2 | 4 | 3
  Erythrocytes; above normal range | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Granular casts; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Granular casts; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Granular casts; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Granular casts; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyaline casts; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Hyaline casts; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyaline casts; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Hyaline casts; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 2 | 4 | 3
  Leukocytes; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocytes; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 2 | 4 | 3
  Leukocytes; above normal range | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
  RBC cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  RBC cast; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  RBC cast; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  WBC cast; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  WBC cast; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Waxy cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Waxy cast; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Waxy cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 2
  Waxy cast; above normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH; below normal range | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH; above normal range | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

66. Primary Outcome: Part B: Number of Participants With Abnormal Urinalysis Results Anytime Between 40 to 48 Hours Post-Dose 10
Description: Following urine parameters were analysed: epithelial cells (normal range: 0 to 5 cells per hpf), erythrocytes (0 to 2 per hpf), granular casts (0 per lpf), hyaline casts (0 to 1 per lpf), leukocytes (0 to 5 per hpf), RBC casts (0 per lpf), WBC casts (0 per lpf), waxy casts (0 per lpf) and pH (5 to 8).
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 5
Participants
  Epithelial Cells; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Epithelial Cells; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Epithelial Cells; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Epithelial Cells; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Erythrocytes; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 2
  Erythrocytes; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Erythrocytes; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 2
  Erythrocytes; above normal range | 0 | 0 | 1 | 0 |  |  | 2 | 0
  Granular casts; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Granular casts; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Granular casts; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Granular casts; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Hyaline casts; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Hyaline casts; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Hyaline casts; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Hyaline casts; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Leukocytes; below normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 2
  Leukocytes; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Leukocytes; above normal range: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 2
  Leukocytes; above normal range | 0 | 0 | 0 | 0 |  |  | 1 | 0
  RBC cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  RBC cast; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  RBC cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  RBC cast; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  WBC cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  WBC cast; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  WBC cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  WBC cast; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Waxy cast; below normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Waxy cast; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  Waxy cast; above normal range: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Waxy cast; above normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  pH; below normal range | 0 | 0 | 0 | 0 |  |  | 0 | 0
  pH; above normal range | 1 | 0 | 1 | 1 |  |  | 0 | 2

67. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Baseline
Description: A 12-lead ECG was performed for assessment of following ECG parameters: ventricular heart rate, PR interval, QRS interval, QT interval and QT interval corrected by Bazzett's formula (QTcB) interval. Number of participants with abnormal clinically significant results for any ECG parameter per investigator's interpretation are reported in this outcome measure.
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants | 0 | 0 | 0 | 0

68. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose
Description: A 12-lead ECG was performed for assessment of following ECG parameters: ventricular heart rate, PR interval, QRS interval, QT interval and QTcB interval. Number of participants with abnormal clinically significant results for any ECG parameter per investigator's interpretation are reported in this outcome measure.
Time Frame: Anytime between 4 to 5 hours post-dose on Day 1
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 7 | 3 | 6
Participants | 0 | 0 | 0 | 0

69. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation Anytime Between 18 to 24 Hours Post-dose
Description: as for outcome 68
Time Frame: Anytime between 18 to 24 hours post-dose on Day 1
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0

70. Primary Outcome: Part A: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at 48 Hours Post-dose
Description: as for outcome 68
Time Frame: 48 hours post-dose on Day 1
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RV521 1.0 mg/kg | Cohort 1: RV521 2.0 mg/kg | Cohort 1: RV521 2.5 mg/kg | Cohort 2: RV521 2.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 2 | 6
Participants | 0 | 1 | 0 | 0

71. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Baseline
Description: as for outcome 68
Time Frame: Baseline (pre-dose on Day 1)
Population: Safety population included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 1 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

72. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose 1
Description: as for outcome 68
Time Frame: Anytime between 4 to 5 hours post-dose 1 on Day 1
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 3 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

73. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Pre-dose 3
Description: as for outcome 68
Time Frame: Pre-dose 3 (Day 2)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

74. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Pre-dose 5
Description: as for outcome 68
Time Frame: Pre-dose 5 (Day 3)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

75. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation Anytime Between 4 to 5 Hours Post-Dose 6
Description: as for outcome 68
Time Frame: Anytime between 4 to 5 hours post-dose 6 (Day 3)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 4 | 4 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

76. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Pre-dose 8
Description: as for outcome 68
Time Frame: Pre-dose 8 (Day 4)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 1 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

77. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation at Pre-dose 10
Description: as for outcome 68
Time Frame: Pre-dose 10 (Day 5)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 1 | 2 | 1 | 0 | 0 | 3 | 3 | 4
Participants | 0 | 0 | 0 |  |  | 0 | 0 | 0

78. Primary Outcome: Part B: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Results Per Investigator's Interpretation Anytime Between 40 to 48 Hours Post-Dose 10
Description: as for outcome 68
Time Frame: Anytime between 40 to 48 hours post-dose 10 on Day 5
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: RSV1 2.5 mg/kg | Cohort 3: RV521 3.5 mg/kg | Cohort 3: RV521 5 mg/kg | Cohort 4: Placebo | Cohort 4: RV521 2.5 mg/kg | Cohort 5: Placebo | Cohort 5: RV521 2.5 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 0 | 4 | 5 | 8
Participants | 0 | 0 | 0 | 0 |  | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of IMP on Day 1 up to Day 7 for Part A; From start of IMP on Day 1 up to Day 12 for Part B
Description: Same event may appear as SAE and non-SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another or 1 participant may have experienced both serious and non-serious event during study. Safety population included all participants who received at least 1 dose of IMP.
Groups:
- Part A: Cohort 1: RV521 1.0 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 1.0 milligram per kilogram (mg/kg) of RV521 orally on Day 1.
- Part A: Cohort 1: RV521 2.0 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 2.0 mg/kg of RV521 orally on Day 1.
- Part A: Cohort 1: RV521 2.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received a single dose of 2.5 mg/kg of RV521 orally on Day 1.
- Part A: Cohort 2: RV521 2.0 mg/kg: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received a single dose of 2 mg/kg of RV521 orally on Day 1.
- Part B: Cohort 3: Placebo: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received placebo every 12 hours twice daily (BID) orally for 5 days.
- Part B: Cohort 3: RSV1 2.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 2.5 mg/kg every 12 hours (BID) orally for 5 days.
- Part B: Cohort 3: RV521 3.5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 3.5 mg/kg every 12 hours (BID) orally for 5 days.
- Part B: Cohort 3: RV521 5 mg/kg: Infants aged >=6 months to <=36 months hospitalized with RSV LRTI received RV521 5 mg/kg every 12 hours (BID) orally for 5 days.
- Part B: Cohort 4: Placebo; Part B: Cohort 5: Placebo: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received placebo every 12 hours (BID) orally for 5 days.
- Part B: Cohort 4: RV521 2.5 mg/kg; Part B: Cohort 5: RV521 2.5 mg/kg: Infants aged >=1 month to <6 months hospitalized with RSV LRTI received RV521 2.5 mg/kg every 12 hours (BID) orally for 5 days.
Arm/Group | Part A: Cohort 1: RV521 1.0 mg/kg | Part A: Cohort 1: RV521 2.0 mg/kg | Part A: Cohort 1: RV521 2.5 mg/kg | Part A: Cohort 2: RV521 2.0 mg/kg | Part B: Cohort 3: Placebo | Part B: Cohort 3: RSV1 2.5 mg/kg | Part B: Cohort 3: RV521 3.5 mg/kg | Part B: Cohort 3: RV521 5 mg/kg | Part B: Cohort 4: Placebo | Part B: Cohort 4: RV521 2.5 mg/kg | Part B: Cohort 5: Placebo | Part B: Cohort 5: RV521 2.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/3 | 0/6 | 0/3 | 0/3 | 0/4 | 0/3 | 0/1 | 0/4 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 0/3 | 0/6 | 0/3 | 0/3 | 0/4 | 0/3 | 0/1 | 0/4 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 2/3 | 4/7 | 3/3 | 1/6 | 1/3 | 2/3 | 1/4 | 1/3 | 1/1 | 2/4 | 3/5 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: RV521 1.0 mg/kg (N=3) | Part A: Cohort 1: RV521 2.0 mg/kg (N=7) | Part A: Cohort 1: RV521 2.5 mg/kg (N=3) | Part A: Cohort 2: RV521 2.0 mg/kg (N=6) | Part B: Cohort 3: Placebo (N=3) | Part B: Cohort 3: RSV1 2.5 mg/kg (N=3) | Part B: Cohort 3: RV521 3.5 mg/kg (N=4) | Part B: Cohort 3: RV521 5 mg/kg (N=3) | Part B: Cohort 4: Placebo (N=1) | Part B: Cohort 4: RV521 2.5 mg/kg (N=4) | Part B: Cohort 5: Placebo (N=5) | Part B: Cohort 5: RV521 2.5 mg/kg (N=8)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1: RV521 1.0 mg/kg (N=3) | Part A: Cohort 1: RV521 2.0 mg/kg (N=7) | Part A: Cohort 1: RV521 2.5 mg/kg (N=3) | Part A: Cohort 2: RV521 2.0 mg/kg (N=6) | Part B: Cohort 3: Placebo (N=3) | Part B: Cohort 3: RSV1 2.5 mg/kg (N=3) | Part B: Cohort 3: RV521 3.5 mg/kg (N=4) | Part B: Cohort 3: RV521 5 mg/kg (N=3) | Part B: Cohort 4: Placebo (N=1) | Part B: Cohort 4: RV521 2.5 mg/kg (N=4) | Part B: Cohort 5: Placebo (N=5) | Part B: Cohort 5: RV521 2.5 mg/kg (N=8)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT04225897/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04225897/SAP_001.pdf